CLINICAL TRIAL: NCT05021952
Title: Effects of Postoperative Prognosis Management Service Using Mobile Applications and Smart Bands for Prostate Cancer Patients
Brief Title: Postoperative Prognosis Management Service Based mHealth for Prostate Cancer Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Seoul St. Mary's Hospital (Other)
Collaborators: National IT Industry Promotion Agency (Unknown)
Responsible Party: Principal Investigator, Ji Youl Lee, Professor, Seoul St. Mary's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: NIPA AIoT_Cancer
Record Dates: First submitted 2021-08-19; First posted 2021-08-26 (Actual); Last update posted 2021-08-26 (Actual); Status verified 2021-08

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Wearable Electronic Devices

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- mHealth App and wearable device (Experimental): An intervention group (App+IoT device) uses a smart care application for 12 months. This application was tailored for prostate cancer patients and created by reflecting the treatment process after surgery. And they also uses a wearable smart band for 12 months.
  Interventions: Device: mHealth App and wearable device
- Education brochure (No Intervention): Control group is provided general education through the hospital brochure.

INTERVENTIONS:
Device: mHealth App and wearable device — An intervention group (App+IoT device) uses a smart care application for 12 months. This application was tailored for prostate cancer patients and created by reflecting the treatment process after surgery. And they also uses a wearable smart band for 12 months.
  Arms: mHealth App and wearable device

SUMMARY:
Recently, the use of mobile health is increasing for the purpose of managing prognosis such as recurrence, survival and quality of life by using a wearable smart band and a smartphone application. In the era of the 4th revolution, mobile health for the purpose of comprehensive prognosis for cancer patients is becoming a very good tool.

It is possible to confirm the clinical significance of short-term and temporary health care through a mobile application and a smart band during the treatment process for cancer patients, but the study is insufficient to generalize the number of subjects.

Therefore, for prostate cancer patients who need prognosis management after surgery, we will investigate the effect of a mobile application using a smart band which has a modular structure reflecting the treatment method and treatment process after surgery.

This study targets patients who underwent prostate cancer surgery. An intervention group (App+IoT device) uses a smart care application for 12 months. This application was tailored for prostate cancer patients and created by reflecting the treatment process after surgery. And they also uses a wearable smart band for 12 months. Control group is provided general education through the hospital brochure. Evaluation will be conducted 2-3days after surgery (before discharge), and at 1, 3, 6, and 12 months after surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients 19 years of age or older who have been diagnosed with prostate cancer
* Patients who have completed surgical treatment for cancer within 3 months of screening and have no additional treatment planned
* Patients who can use a prognosis management application and can perform regular follow-up examinations in outpatient settings
* Patients carrying an Android or iOS smartphone
* Patients who voluntarily decide to participate and give written consent after hearing detailed explanations about this study

Exclusion Criteria:

* Patients who have been treated within the last 3 months for other serious diseases (hematologic cancer, malignancy, etc.)
* Patients for whom additional treatment was planned due to cancer recurrence or metastasis
* Patients with severe cardiopulmonary disease who are unable to proceed with rehabilitation exercise programs
* Patients who find it difficult to proceed with the rehabilitation exercise program due to pain caused by bone metastasis and concerns about pathological fractures
* Patients who underwent lower extremity artificial joint TKRA and THRA
* Patients who are not eligible for rehabilitation exercise as judged by medical personnel

Ages: 19 Years to 100 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 324 (Estimated)
Dates: Start 2021-05-21 (Actual); Primary Completion 2023-05-30 (Estimated); Study Completion 2024-05-30 (Estimated)

PRIMARY OUTCOMES:
Change of body composition (weight, kg) | Enrollment (postoperative 2-3days), postoperative 1month, 3month, 6month, 12month
  According to time frame with between-group and within group, trends will be found.

SECONDARY OUTCOMES:
Change of Quality of life (EORTC-QLQ-C30) | Enrollment (postoperative 2-3days), postoperative 1month, 3month, 6month, 12month
  According to time frame with between-group and within group, trends will be found.
  This questionnaire contains 30 items regarding general health status, five functional scales (ie, physical, role, cognitive, emotional, and social functioning), three symptom scales (ie, fatigue, pain, and nausea or vomiting), and six single-item scales (ie, dyspnea, appetite loss, constipation, diarrhea, financial difficulties, and insomnia).
Pain (Numeric rating scale, NRS) | Enrollment (postoperative 2-3days), postoperative 1month, 3month, 6month, 12month
  According to time frame with between-group and within group, trends will be found. NRS score (11 point scales) ranges from 0 (no pain) to 10 (possible to image maximum pain). A higher score means more pain.
Self-reported symptom and Quality of life (EORTC-QLQ-PR25) | Enrollment (postoperative 2-3days), postoperative 1month, 3month, 6month, 12month
  According to time frame with between-group and within group, trends will be found. EORTC-QLQ-PR25 consists of 25 questions and identifies various symptoms or problems that patients may experience.
Physical activity (IPAQ-SF) | Enrollment (postoperative 2-3days), postoperative 1month, 3month, 6month, 12month
  According to time frame with between-group and within group, trends will be found. IPAQ-SF finds out about the physical activities that patients do on a daily basis. This includes activities that patients do at work or at home, activities they do while using transportation, activities they do in their spare time, and exercise. This questionnaire consists of 7 questions.
Urination Symptom (ICIQ-SF) | Enrollment (postoperative 2-3days), postoperative 1month, 3month, 6month, 12month
  According to time frame with between-group and within group, trends will be found. ICIQ-SF is about the urine symptom that patients are experiencing, and consists of a total of 4 questions.
Overactive Bladder Symptom (OABSS) | Enrollment (postoperative 2-3days), postoperative 1month, 3month, 6month, 12month
  According to time frame with between-group and within group, trends will be found. OABSS is a questionnaire about overactive bladder symptom and consists of a total of 4 items.
Prostatic Hyperplasia (IPSS) | Enrollment (postoperative 2-3days), postoperative 1month, 3month, 6month, 12month
  According to time frame with between-group and within group, trends will be found. IPSS is a questionnaire about prostatic hyperplasia to find out uncomfortable symptoms that may appear when urinating. This questionnaire consists of 8 questions.
Erectile Dysfunction Symptom (IIEF-5) | Enrollment (postoperative 2-3days), postoperative 1month, 3month, 6month, 12month
  According to time frame with between-group and within group, trends will be found. IIEF-5 is a questionnaire about the symptoms of erectile dysfunction that may appear after surgery, and consists of 5 questions.
Grip strength | Enrollment (postoperative 2-3days), postoperative 1month, 3month, 6month, 12month
  According to time frame with between-group and within group, trends will be found. Using a grip dynamometer, take three measurements on both hands. Higher value (kg) indicates higher grip strength.
Lower extremity muscle endurance (30seconds chair stands test) | Enrollment (postoperative 2-3days), postoperative 1month, 3month, 6month, 12month
  According to time frame with between-group and within group, trends will be found. It measures the number of times you sit down and stand up from a chair in 30 seconds. Higher value (number) indicates higher lower extremity muscle endurance.
  It is judged that the 30seconds chair stands test will be difficult due to abdominal pain after surgery, so the evaluation is performed only at the other F/U points excluding the enrollment date.
2 Minute walk test (2MWT, evaluation of cardiopulmonary endurance) | Enrollment (postoperative 2-3days), postoperative 1month, 3month, 6month, 12month
  According to time frame with between-group and within group, trends will be found. The 2MWT is a measurement of endurance that assesses walking distance over two minutes.
  It is judged that the 2MWT will be difficult due to abdominal pain after surgery, so the evaluation is performed only at the other F/U points excluding the enrollment date.
Nutrition assessment (Mini-nutrition assessment, MNA) | Enrollment (postoperative 2-3days), postoperative 1month, 3month, 6month, 12month
  According to time frame with between-group and within group, trends will be found. The short form of the MNA (MNASF) is a screening tool consisting of six questions on food intake, weight loss, mobility, psychological stress, or acute disease, the presence of dementia or depression, and body mass index (BMI). The maximum score for this part is equal to 14. A score equal to or higher than 12 indicates that the subject under study has an acceptable nutritional status thus excluding malnutrition and/or malnutrition risk, meanwhile, a score ≤ 11 implicates to proceed with the complete version of the MNA (MNA-LF). This version consists of 12 additional items and provides a maximum possible overall assessment of 30 scores: a score of fewer than 17 indicates malnutrition, a score of 17-23.5 indicates a risk for malnutrition and a score higher 23.5 indicates well-nourishment.

CONTACTS AND LOCATIONS:
Overall Officials: JIYOUL LEE, Professor, Principal Investigator — Department of Urology Seoul St. Mary's Hospital
Locations (1):
- Korea University Anam Hospital, Seoul, Seongbuk-gu, South Korea

IPD SHARING:
Plan to Share IPD: No